CLINICAL TRIAL: NCT01833637
Title: Electronic Patient Reported Symptom Assessment: A Pilot Study Introducing Advanced Care Planning and Palliative Care to Hospitalized Women With Advanced Gynecologic, Breast, Thoracic, or Gastrointestinal Malignancies.
Brief Title: Electronic Patient Reported Symptom Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emily Berry, Physician, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00064629
Record Dates: First submitted 2012-10-23; First posted 2013-04-17 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Gynecologic Cancer; Breast Cancer; Thoracic Cancer; Gastrointestinal Cancer
Keywords: Advanced Care Planning; Palliative Care; Women
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Control Group (No Intervention): Patients randomized to the control group will be asked to fill out a patient symptom questionnaire using an iPad at the time of registration and then every 24 hours until released from the hospital. It should take about 10 minutes to complete the questions each time. The survey will not interfere with the care the healthcare team will be providing. Patients will be asked to fill our a Patient Satisfaction Questionnaire at the time of discharge.
- Arm B: APN Intervention Group (Active Comparator): Patients randomized to this group will be asked to fill out a patient symptom assessment using an iPad at the time of registration and then every day until released from the hospital. It should take about 10 minutes to complete this questionnaire each time. Based on the patients' answers and in cooperation with their health care provider, an Advanced Practice Nurse (APN) will provide information about symptom management and options for services that are available after the patient leaves the hospital. The survey responses will be shared with the patients' healthcare team so that they better understand how they are feeling. The APN will work closely with the healthcare team. Patients will be asked to fill out a Patient Satisfaction Questionnaire at the time of discharge.
  Interventions: Other: APN Intervention

INTERVENTIONS:
Other: APN Intervention — Patients randomized to this group will be asked to fill out a patient symptom assessment using an iPad at the time of registration and then every day until released from the hospital. It should take about 10 minutes to complete this questionnaire each time. Based on the patients' answers and in cooperation with their health care provider, an Advanced Practice Nurse (APN) will provide information about symptom management and options for services that are available after the patient leaves the hospital. The survey responses will be shared with the patients' healthcare team so that they better understand how they are feeling. The APN will work closely with the healthcare team. Patients will be asked to fill out a Patient Satisfaction Questionnaire at the time of discharge.
  Arms: Arm B: APN Intervention Group

SUMMARY:
The purpose of this study is to assess whether using computerized screening questions can improve how well we manage symptoms related to cancer and cancer treatments. Advance care planning is a process in which teams of experts assist in with treatment plans, managing pain and other symptoms, emotional issues, and end of life issues. With advances in technology, it is now possible to get the patient's feedback directly and more often. It is thought that repeated questionnaires completed by the patient will provide a better and more accurate measure of the patient's needs and experiences but this has not been tested. This study is designed to learn if using a computerized assessment repeatedly is better than standard planning techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have a diagnosis of metastatic breast, gynecologic, thoracic, or gastrointestinal malignancy. Women diagnosed with non-solid organ tumors (i.e., lymphoma, leukemia) will be excluded as their symptom profile in advanced/metastatic disease is dissimilar.
2. Reason for admission must be for symptom management from cancer or cancer therapy.
3. Patients must be age 18 or older.
4. Only patients cared for at the Robert H. Lurie Comprehensive Cancer Center (RHLCCC) will be eligible for this small pilot study.
5. Patients must not be enrolled in hospice care.
6. Patients must have a performance status 0-3 (ECOG scale).
7. Patients must be alert and oriented to time, place, and person. Must be able to answer questions.
8. Patients must be able to speak, read, and communicate in English.
9. Patients must have a signed consent and authorization for research and be amenable to be followed for outcomes/response throughout and after hospitalization.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Identify perceived symptom burden and quality of life in our female patients with advanced gynecologic, breast, thoracic, or gastrointestinal malignancies. | 3 years
  We will compare the symptom scores of the control and the intervention groups to determine if the overall symptom burden scores are lower and patient satisfaction scores are higher in the group who receive targeted intervention combined with education.
Trend perceived symptom burden and quality of life in our female patients with advanced gynecologic, breast, thoracic, or gastrointestinal malignancies. | 3 years
  We will compare the symptom scores of the control and the intervention groups to determine if the overall symptom burden scores are lower and patient satisfaction scores are higher in the group who receive targeted intervention combined with education.

SECONDARY OUTCOMES:
Examine scores of electronic reported symptom assessment combined with targeted intervention to see it it improves symptoms scores over the course of hospitalization. | 3 years
Use electronic symptom scoring, targeted intervention, and sequential assessments every 24 hours to assess the impact on length of hospitalization and readmissions. | 3 years
Assess level of understanding about advance care planning in both the control and intervention group. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily Berry, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States